CLINICAL TRIAL: NCT05965232
Title: Screening for Severe Hepatic Fibrosis by FibroScan in a Population Presenting a Severe Psychiatric Disorder Under Treatment for at Least Two Years.
Brief Title: FIbrosis and Steatosis in Patients With Psychiatric Illness
Acronym: FibroPsy
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Esquirol (Other)
Responsible Party: Principal Investigator, Philippe Nubukpo, Professor, Centre Hospitalier Esquirol
Other Study IDs: 2017-A01998-45
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Severe Bipolar I Disorder (Diagnosis); Bipolar I Disorder, Most Recent Episode Mixed, in Remission; Depression Psychotic Feature; Mood-Incongruent Delusion
MeSH Terms: conditions — Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1 dry tube to obtain serum (7 mL) and one heparinized tube for whole blood (7 mL) will be collected
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fibroscan — Performing FibroScan :
  The patient is positioned supine, with the right arm in maximum abduction to clear the intercostal spaces.The measurement itself is performed on the right lobe of the liver via the intercostal (intersection of the mid-axillary line and the xiphoid process) using a dedicated probe (3.5 MHz) after application of a conduction gel to the skin. FibroScan® examinations are carried out by personnel trained in the use of the device.This training is specific and validated by the device's manufacturer manufacturer, EchosensTM (Paris). Ten valid measurements at the same measurement point in the right liver must be be performed, with an interquartile range/median ratio ≤ 30 (required only if the elastometry value is > 7.1 KPa.
  Other Names: Blood sample

SUMMARY:
Background: Severe psychiatric diseases (schizophrenia, bipolarity, depression, anxious syndrome) are often associated with a metabolic syndrome, including Non-Alcoholic Steato Hepatitis, probably misdiagnosed in patients with psychiatric illness. Furthermore, long-term exposition to substances like alcohol or to one or more psychotropic treatments may involve liver detoxification role. Thanks to liver stiffness, based on FibroScan®, and CAP (controlled attenuation parameter), we wanted to study prevalence of severe fibrosis and steatosis in this population.

Material & Methods: Prospective study of 385 subjects hospitalised in a psychiatric hospital for schizophrenia, bipolar disorder, depression or anxiety-depression disorder and receiving psychotropic treatment for at least 2 years, for whom a FibroScan®, a blood test and a record of clinical data were carried out, after information and informed consent.

Benefits expected : This study should show an expected excess risk of fibrosis. FibroScan® in this population and determine the risk factors more associated risk factors. Generalized or targeted screening for identified risk factors in this population could help optimize in this population could help optimize the choice and dosage of psychotropic of psychotropic drugs, and above all, help to guide the strategy of hepatic and prevention strategy.

DETAILED DESCRIPTION:
Patients with psychiatric illness are often exposed to an increase risk of mortality compared to the general population: a reduction of life expectancy between 7 and 24 years has been described . Somatic illnesses explain 60% of this excess of mortality, particularly cardiovascular diseases . Notably, patients with chronic psychiatric disorders, such as depression, bipolar disorders or schizophrenia are more frequently exposed to metabolic syndrome. A recent meta-analysis showed that patients with severe mental illness had a RR of 1.58 (1.35-1.86) of developing metabolic syndrome.

Steatosis, or fat excess in hepatocytes defines NAFLD (non-alcoholic fatty liver disease). NAFLD is a spectrum of liver illnesses associated with metabolic syndrome. Within NAFLD, NASH (non-alcoholic steatohepatitis) occurs in about 5 % of the cases, liver inflammation and/or fibrosis being associated to steatosis: Survival is then impaired, notably with a specific risk of cirrhosis in 20% of the patients with NASH and 3 % of patients with NAFLD . Hepatocarcinoma is a complication of cirrhosis but it may be observed in the absence of cirrhosis in nearly 30% of the cases. Its prevalence is progressively increasing, from 20 to 27%. It will probably be the leading cause of liver transplantation in the next years Otherwise, patients with NAFLD are also exposed to non-liver related complications: cardiovascular risk is higher in this population and is the main risk of mortality.

Although NAFLD is a frequent disease, it is yet generally misdiagnosed today, essentially because of the lack of symptoms and of systematic screening. Furthermore, it is key to diagnose the evolutionary stage: pure NAFLD, NASH and stage of fibrosis. The liver biopsy remains the gold standard, despite its limitations linked to the sample variability and the differences in interpretation even between expert pathologists.

However, specific risks associated with this procedure, such as bleeding and even a marginal risk of death have been described. Furthermore, liver biopsy is costly. All these arguments explain the difficulty to apply this invasive strategy in screening in the general population. That's why different methods, based on non-invasive tests, were developed to diagnose fibrosis - the main prognostic factor - and more recently in a more preliminary way to assess steatosis and inflammation. Two main methods are used to evaluate fibrosis stage: serum biomarkers and liver stiffness. Serum biomarkers are non-parametric (for example NAFLD fibrosis score, Fib4, Forns score and more recently, eLIFT.) or parametric (for example FibroTest, FibroMeter.). Liver stiffness is mainly assessed by FibroScan: it is easily available, and reproducible. It was largely validated in different liver diseases, including NAFLD. Steatosis is simultaneously evaluated, thanks to CAP (controlled attenuation parameter.). Strategies based on the associations of different markers have been evaluated to increase sensibility and specificity of each method taken alone to assess fibrosis. Specific combinations of elastometry and biomarkers have emerged, such as FibroMeterVCTE, and FAST.

In the psychiatric field, NAFLD screening may be important to help to identify patients at liver risk and also at a potential metabolic risk especially since a specific management is available.

Even if the association between NAFLD and psychiatric disorders has been described, its exact prevalence and impact are not well identified.

This is why we aimed to explore the prevalence of liver fibrosis and steatosis in patients with chronic psychiatric illnesses. We led a prospective descriptive single-center study in the Esquirol psychiatric hospital in Limoges.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a severe psychiatric disorder (psychotic disorder, mood disorder, anxiety or anxiety disorder), and under psychotropic treatment (neuroleptic and/or antidepressant) for at least two years.

and/or antidepressant) for at least two years, and hospitalized in units treating these disorders in the investigating centers.

- Subjects or their legal representatives who have given informed consent, with social insurance, aged over 18 years of age.

Exclusion Criteria:

* Short-term life-threatening conditions
* Liver disease already diagnosed at inclusion: cancer, cirrhosis, chronic or acute or acute liver disease
* No antipsychotic or antidepressant treatment
* Anti-viral treatment demonstrating infection with hepatitis viruses or the HIV virus (or known positive HIV serology)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects hospitalised in a psychiatric hospital for schizophrenia, bipolar disorder, depression or anxiety-depression disorder and receiving psychotropic treatment for at least 2 years,
Sampling Method: Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-02-08 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Severe fibrosis assessed by FibroScan® in the population of subjects with a severe psychiatric disorder who have been on psychotropic medication for more than than two years | one day
  The cut-off selected for FibroScan® ≥ 8.7 kPa is that published for the diagnosis of severe fibrosis. It is considered clinically relevant associated with a poorer prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe B NUBUKPO, PhD, Principal Investigator — Centre Hospitalier Esquirol
Locations (1):
- Centre Hospitalier Esquirol, Limoges, France